CLINICAL TRIAL: NCT04878211
Title: An Open-label Multicenter Study to Assess Response to COVID-19 Vaccine in Participants With Multiple Sclerosis Treated With Ofatumumab 20 mg Subcutaneously
Brief Title: A Open-label Study to Assess Response to COVID-19 Vaccine in Multiple Sclerosis Participants Treated With Ofatumumab
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Trial was terminated for business reasons. There has been no change in the benefit/risk profile of ofatumumab.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMB157GUS16
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Relapsing Multiple Sclerosis (RMS)
Keywords: Multiple Sclerosis; Relapsing Multiple Sclerosis; COVID; COVID-19; Vaccine; Coronavirus; adult; OMB157
MeSH Terms: conditions — Multiple Sclerosis; COVID-19; Coronavirus Infections | interventions — ofatumumab; CVnCoV COVID-19 vaccine; Interferons; Glatiramer Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 - 2 WKs vaccine prior to OMB157 (Experimental): Participants received non-live COVID-19 mRNA vaccine at least two weeks prior to start of ofatumumab (OMB157) (20 mg subcutaneous).
  Interventions: Drug: Ofatumumab; Biological: mRNA COVID-19 vaccine
- Cohort 2 - vaccine 4 WKs after OMB157 (Experimental): Participants received non-live COVID-19 mRNA vaccine at least four weeks after start of ofatumumab (OMB157) (20 mg subcutaneous).
  Interventions: Drug: Ofatumumab; Biological: mRNA COVID-19 vaccine
- Cohort 3 - Interferon or glatiramer acetate - vaccine 4 WKs after (Active Comparator): Participants will receive non-live COVID-19 mRNA vaccine at least 4 weeks after start of prescribed interferon or glatiramer acetate
  Interventions: Biological: mRNA COVID-19 vaccine; Drug: interferon or glatiramer acetate
- Cohort 4 - Fully vaccinated and on OMB457 ≥ 4 WKs (Experimental): Participants fully vaccinated with a non-live COVID mRNA vaccine and on ofatumumab for at least 4 weeks (20 mg subcutaneous)
  Interventions: Drug: Ofatumumab; Biological: mRNA COVID-19 vaccine
- Cohort 5 -Fully vaccinated, on interferon or glatiramer acetate for ≥ 4 WKs ± booster (Experimental): Participants fully vaccinated with a non-live COVID mRNA vaccine, without or without a booster, and on interferon or glatiramer acetate for at least 4 weeks.
  Interventions: Biological: mRNA COVID-19 vaccine; Drug: interferon or glatiramer acetate
- Cohort 6 - Fully vaccinated, currently on OMB457 for ≥ 4 WKs, + booster (Experimental): Participants fully vaccinated with a non-live COVID mRNA vaccine with a booster and on ofatumumab for at least 4 weeks (20 mg subcutaneous)
  Interventions: Drug: Ofatumumab; Biological: mRNA COVID-19 vaccine

INTERVENTIONS:
Drug: Ofatumumab — 3 loading doses followed by monthly administrations
  Arms: Cohort 1 - 2 WKs vaccine prior to OMB157; Cohort 2 - vaccine 4 WKs after OMB157; Cohort 4 - Fully vaccinated and on OMB457 ≥ 4 WKs; Cohort 6 - Fully vaccinated, currently on OMB457 for ≥ 4 WKs, + booster
Biological: mRNA COVID-19 vaccine — Pfizer or Moderna mRNA Vaccine
Drug: interferon or glatiramer acetate — iDMT
  Arms: Cohort 3 - Interferon or glatiramer acetate - vaccine 4 WKs after; Cohort 5 -Fully vaccinated, on interferon or glatiramer acetate for ≥ 4 WKs ± booster

SUMMARY:
This study evaluated if relapsing multiple sclerosis (MS) participants treated with ofatumumab 20 mg subcutaneous (s.c.) administered once monthly could develop an adequate immune response to the COVID-19 mRNA vaccine compared to participants on an interferon or glatiramer acetate.

DETAILED DESCRIPTION:
This was a six-cohort, multicenter, prospective study planned for up to 88 relapsing multiple sclerosis (MS) participants. The study was intended to address two questions: 1) Can participants treated with ofatumumab develop an immune response if receiving a COVID-19 mRNA vaccine two weeks prior to ofatumumab start? 2) If receiving COVID-19 mRNA vaccine after introduction of ofatumumab treatment, can participants develop an immune response? Cohort 1: participants received an mRNA COVID-19 vaccine at least two weeks prior to ofatumumab start. Cohort 2: participants received an mRNA COVID-19 vaccine at least four weeks after beginning ofatumumab. Cohort 3: participants on an interferon or glatiramer acetate who received COVID-19 mRNA vaccine. Cohort 4: participants fully vaccinated with an RNA COVID-19 vaccine at least four weeks after ofatumumab start. Cohort 5: participants vaccinated with an RNA COVID-19 vaccine, with or without a booster dose, and on interferon or glatiramer acetate. Cohort 6: participants fully vaccinated with an RNA COVID-19 vaccine who received a booster dose at least four weeks after ofatumumab start. Participants obtained the COVID-19 mRNA vaccine from their HCP (private insurance) or appropriate federal, state or local program.

Participants in Cohort 1 received loading doses of ofatumumab and subsequent dosing was 20 mg s.c. administered monthly. All other cohorts continued current dosing schedule of either ofatumumab, glatiramer acetate or interferon. Participation in trial was maximum of 421 days which was dependent on the Cohort.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Diagnosis of relapsing MS by 2017 revised McDonald criteria
* Were willing to comply with the study schedule
* Cohort 1: Were receiving an mRNA COVID-19 vaccine (Pfizer or Moderna vaccine) at least two weeks prior to starting ofatumumab
* Cohort 2: Were receiving an mRNA COVID-19 vaccine (Pfizer or Moderna vaccine) and on ofatumumab for at least 4 weeks
* Cohort 3: Were receiving an mRNA COVID-19 vaccine (Pfizer or Moderna vaccine) and on interferon or glatiramer acetate for at least 4 weeks
* Cohort 4: Fully vaccinated with a non-live COVID mRNA vaccine (Pfizer or Moderna vaccine) and on ofatumumab for at least 4 weeks
* Cohort 5: Fully vaccinated with a non-live COVID mRNA vaccine (Pfizer or Moderna vaccine), with or without a booster, and on interferon or glatiramer acetate for at least 4 weeks
* Cohort 6: Fully vaccinated with a non-live COVID mRNA vaccine, (Pfizer or Moderna vaccine), with a booster, and on ofatumumab for at least 4 weeks

Exclusion Criteria:

* Received the J&J vaccine.
* Had a contraindication to receiving an mRNA COVID-19 vaccine
* Had an immediate allergic reaction to past vaccine or injection
* Experienced a major episode of infection requiring hospitalization or treatment with intravenous antibiotics within 2 weeks prior to the screening visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Center For Neurology and Spine, Phoenix, Arizona
  - Infinity Clinical Research LLC ., Hollywood, Florida
  - Dragonfly Research LLC, Wellesley, Massachusetts
  - Minnesota Center Multiple Sclerosis, Plymouth, Minnesota
  - The MS Center for Innovation in Care, St Louis, Missouri
  - The Neurological Institute PA, Charlotte, North Carolina
  - Dayton Center for Neurological Disorders, Centerville, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2308

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 24 participants screened.
  Cohort = C
Groups:
- C1: VN - Plan to Start OMB157: Vaccine naive, planning to start ofatumumab
- C2: VN - on OMB157 >=4 WKs: Vaccine naive, currently on ofatumumab for ≥ 4 weeks
- C3: VN - INFy or GA >=4 WKs: Vaccine naive, on interferon or glatiramer acetate for ≥ 4 weeks
- C4: FV - OMB157 >=4 WKs: Fully vaccinated, currently on ofatumumab for ≥ 4 weeks
- C5: FV - INFy or GA >=4 WKs: Fully vaccinated, on interferon or glatiramer acetate for ≥ 4 weeks
- C6: FV - on OMB157 >=4 WKs + Booster: Fully vaccinated, currently on ofatumumab for ≥ 4 weeks,
  + booster
Period: Overall Study
Arm/Group | C1: VN - Plan to Start OMB157 | C2: VN - on OMB157 >=4 WKs | C3: VN - INFy or GA >=4 WKs | C4: FV - OMB157 >=4 WKs | C5: FV - INFy or GA >=4 WKs | C6: FV - on OMB157 >=4 WKs + Booster
Started | 5 | 2 | 0 | 1 | 11 | 5
Completed | 4 | 2 | 0 | 0 | 1 | 0
Not Completed | 1 | 0 | 0 | 1 | 10 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Protocol deviation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 9 | 4
Not completed — Subject decision | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: There were no participants enrolled in Cohort 3.
Groups:
- Total: Total of all reporting groups
Arm/Group | C1: VN - Plan to Start OMB157 | C2: VN - on OMB157 >=4 WKs | C3: VN - INFy or GA >=4 WKs | C4: FV - OMB157 >=4 WKs | C5: FV - INFy or GA >=4 WKs | C6: FV - on OMB157 >=4 WKs + Booster | Total
Number analyzed (Participants) | 5 | 2 | 0 | 1 | 11 | 5 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 0 | 1 | 11 | 5 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 0 | 0 | 8 | 5 | 19
  Male | 0 | 1 | 0 | 1 | 3 | 0 | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 3 | 2 |  | 1 | 10 | 4 | 20
  Black or African American | 2 | 0 |  | 0 | 1 | 0 | 3
  Missing | 0 | 0 |  | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Response by SARS-CoV-2 Qualitative IgG Antibody Assay at 14 Days Post-vaccination by Cohort Group and Overall, Non-response Imputation Approach (Safety Analysis Set)
Description: An immune response is defined as a positive SARS-CoV-2 qualitative IgG antibody assay ≥14 days after full course [2 doses] vaccination to non live mRNA COVID-19 vaccine, Participants with a negative or borderline result were considered non-responders, as well as participants with a missing or invalid immune response assessment at 14 days post-vaccination (imputed as non-responders).
Time Frame: Cohorts 1 - 3: >=14 days after vaccination: Day 36 (Pfizer) or Day 43 (Moderna); Cohorts 4-6: Day 1
Population: Safety analysis set (excluding 2 participants diagnosed with COVID-19 prior to study entry. Overall number analyzed included participants who received full course of vaccine (2 doses. n =number of participants with a positive result (responders). M = number of participants in the safety analysis set who received full course (2 doses) of a COVID 19 vaccine, including a COVID-19 booster for Cohort 6 participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Overall: All cohorts
Arm/Group | C1: VN - Plan to Start OMB157 | C2: VN - on OMB157 >=4 WKs | C3: VN - INFy or GA >=4 WKs | C4: FV - OMB157 >=4 WKs | C5: FV - INFy or GA >=4 WKs | C6: FV - on OMB157 >=4 WKs + Booster | Overall
Number analyzed (Participants) | 5 | 2 | 0 | 1 | 11 | 5 | 24
Percentage of participants | 100.0 [47.8 to 100.0] | 100.0 [15.8 to 100.0] |  | 0.0 [0.0 to 97.5] | 100.0 [69.2 to 100.0] | 50.0 [6.8 to 93.2] | 86.4 [65.1 to 97.1]

2. Secondary Outcome: Percentage of Patients With an Immune Response by SARS-CoV-2 Qualitative IgG Antibody Assay by Time Point, Cohort Group and Overall, Non-response Imputation Approach (Safety Analysis Set)
Description: as for outcome 1
Time Frame: Vaccination up to 70, 180, 270 and 360 days
Population: Safety analysis set (excluding 2 participants diagnosed with COVID-19 prior to study entry)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | C1: VN - Plan to Start OMB157 | C2: VN - on OMB157 >=4 WKs | C3: VN - INFy or GA >=4 WKs | C4: FV - OMB157 >=4 WKs | C5: FV - INFy or GA >=4 WKs | C6: FV - on OMB157 >=4 WKs + Booster | Overall
Number analyzed (Participants) | 5 | 2 | 0 | 1 | 11 | 5 | 24
Percentage of participants
  70 days post-vaccination n=5,0,0,0,0,0,5: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 5
  70 days post-vaccination n=5,0,0,0,0,0,5 | 100.0 [47.8 to 100.0] |  |  |  |  |  | 100.0 [47.8 to 100.0]
  180 days post-vaccination, n=5,2,0,1,10,4,22: number analyzed (Participants) | 5 | 2 | 0 | 1 | 10 | 4 | 22
  180 days post-vaccination, n=5,2,0,1,10,4,22 | 80.0 [28.4 to 99.5] | 0.0 [0.0 to 84.2] |  | 100.0 [2.5 to 100.0] | 90.0 [55.5 to 99.7] | 25.0 [0.6 to 80.6] | 68.2 [45.1 to 86.1]
  270 days post-vaccination n=5,2,0,1,10,4,22: number analyzed (Participants) | 5 | 2 | 0 | 1 | 10 | 4 | 22
  270 days post-vaccination n=5,2,0,1,10,4,22 | 60.0 [14.7 to 94.7] | 0.0 [0.0 to 70.8] |  | 0.0 [0.0 to 97.5] | 60.0 [26.2 to 87.8] | 50.0 [6.8 to 93.2] | 50.0 [28.2 to 71.8]
  360 days post-vaccination n=5,2,0,1, 10, 4,22: number analyzed (Participants) | 5 | 2 | 0 | 1 | 10 | 4 | 22
  360 days post-vaccination n=5,2,0,1, 10, 4,22 | 60.0 [14.7 to 94.7] | 0.0 [0.0 to 84.2] |  | 0.0 [0.0 to 97.5] | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 60.2] | 18.2 [5.2 to 40.3]

3. Secondary Outcome: Percentage of Participants Achieving Immune Conversion by Individual Cohort Group and Overall, Non-response Imputation Approach (Safety Analysis Set)
Description: Immune conversion was defined as (i) pre-vaccination absence of SARS-CoV-2 qualitative IgG antibody with any post-vaccination positive SARS-CoV-2 qualitative IgG antibody assay (Cohorts 1-3 only); or (ii) pre vaccination presence of SARS-CoV-2 quantitative IgG antibody (i.e., pre vaccination value ≥0.80 U/mL) with any post-vaccination ≥4-fold increase in SARS-CoV-2 quantitative IgG antibody titer (Cohorts 1-3 only); or (iii) initial negative SARS-CoV-2 nucleocapsid antibody assay with any post-vaccination positive SARS-CoV-2 qualitative IgG antibody assay (Cohorts 4 and 5 only). There was no baseline for Cohort 6 because there was no blood collection prior to vaccination.
Time Frame: Cohorts 1 - 3: >=14 days after vaccination: Day 36 (Pfizer) or Day 43 (Moderna); Cohorts 4-5: Day 1
Population: Safety analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Overall: Includes all cohorts
Arm/Group | C1: VN - Plan to Start OMB157 | C2: VN - on OMB157 >=4 WKs | C3: VN - INFy or GA >=4 WKs | C4: FV - OMB157 >=4 WKs | C5: FV - INFy or GA >=4 WKs | Overall
Number analyzed (Participants) | 5 | 2 | 0 | 1 | 11 | 19
Percentage of participants
  Pre-vac absence and post vac positive n=5,2, 0,0,0,7: number analyzed (Participants) | 5 | 2 | 0 | 0 | 0 | 7
  Pre-vac absence and post vac positive n=5,2, 0,0,0,7 | 80.0 [28.4 to 99.5] | 50.0 [1.3 to 98.7] |  |  |  | 71.4 [29.0 to 96.3]
  Pre-vac presence and post vac ≥4-fold increase n=5,2,0,0,0,7: number analyzed (Participants) | 5 | 2 | 0 | 0 | 0 | 7
  Pre-vac presence and post vac ≥4-fold increase n=5,2,0,0,0,7 | 0 [0.0 to 52.2] | 0.0 [0.0 to 84.2] |  |  |  | 0.0 [0.0 to 41.0]
  Initial negative SARS nucleocapsid with post-vac positive SARS n=0,0,0,1,1,2: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 2
  Initial negative SARS nucleocapsid with post-vac positive SARS n=0,0,0,1,1,2 |  |  |  | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 84.2]
  Immune conversion n=5,2,0,1,1,9: number analyzed (Participants) | 5 | 2 | 0 | 1 | 1 | 9
  Immune conversion n=5,2,0,1,1,9 | 80.0 [28.4 to 99.5] | 50.0 [1.3 to 98.7] |  | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5] | 55.6 [21.2 to 86.3]

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were presented from first day of screening , treatment and 30 day safety follow up to a maximum duration of 421 days.
Description: Cohorts 2 and 4 have been combined as participants were on ofatumumab >4 weeks and Cohort 3 and 5 were combined because both cohorts were on glatiramer acetate or IFN for >4 weeks. Purpose of the trial was to determine if ofatumumab affected immune response.
Groups:
- Cohort 1: C1: VN - plan to start OMB157 Vaccine naive, planning to start ofatumumab
- Cohort 2: C2: VN - on OMB157 >=4 WKs Vaccine naive, currently on ofatumumab for ≥ 4 weeks
- Cohort 3: C3: VN - INFy or GA >=4 WKs Vaccine naive, on interferon or glatiramer acetate for ≥ 4 weeks
- Cohort 4: C4: FV - OMB157 >=4 WKs Fully vaccinated, currently on ofatumumab for ≥ 4 weeks
- Cohort 5: C5: FV - INFy or GA >=4 WKs Fully vaccinated, on interferon or glatiramer acetate for ≥ 4 weeks
- Cohort 6: C6: FV - on OMB157 >=4 WKs + booster Fully vaccinated, currently on ofatumumab for ≥ 4 weeks,
  + booster
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2 | 0/0 | 0/1 | 0/11 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/0 | 0/1 | 1/11 | 1/5
Other Adverse Events (participants affected / at risk) | 5/5 | 1/2 | 0/0 | 0/1 | 2/11 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=2) | Cohort 3 (N=0) | Cohort 4 (N=1) | Cohort 5 (N=11) | Cohort 6 (N=5)
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=2) | Cohort 3 (N=0) | Cohort 4 (N=1) | Cohort 5 (N=11) | Cohort 6 (N=5)
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Influenza A virus test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT04878211/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT04878211/SAP_001.pdf